CLINICAL TRIAL: NCT05059379
Title: A Multicenter Randomized Controlled Phase III Study of Medial vs. Entire Supraclavicualr Lymph Node Radiation Therapy for Patients With Pathologically Positive Axillary Lymph Node and High Risk of Recurrence After Breast Cancer Surgery
Brief Title: Medial vs. Entire Supraclavicular Lymph Node Radiation Therapy for Patients With Invasive Breast Cancer
Acronym: SUCLANODE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The First Affiliated Hospital of University of Science and Technology of China (Other); Quanzhou First Hospital (Other); Jiangyin People's Hospital (Other); Affiliated Hospital of Jiangnan University (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC017
Record Dates: First submitted 2021-09-10; First posted 2021-09-28 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Radiotherapy; Complications; Effect of Radiation Therapy
Keywords: breast cancer; supraclavicular lymph node; radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast/chest wall+undisseted axillary+IMN+medial SCL ( medial SCL radiation) (Active Comparator): Radiation is delivered to the breast/chest wall, undissected axilla, internal mammary nodes and medial supraclavicular node. Treatment will be given by normfractionated or hypofractionated radiotherapy (50Gy/25Fx/5w or 42.5Gy/16Fx/3.5w). IMRT and VMAT technique are recommended.
  Interventions: Radiation: Medial supraclavicular lymph node radiotherapy
- Breast/chest wall+undisseted axillary+IMN+entie SCL (entire SCL radiation) (Experimental): Radiation is delivered to the breast/chest wall, undissected axilla, internal mammary nodes and entire supraclavicular node. Treatment will be given by normfractionated or hypofractionated radiotherapy (50Gy/25Fx/5w or 42.5Gy/16Fx/3.5w). IMRT and VMAT technique are recommended.
  Interventions: Radiation: Entire supraclavicular lymph node radiotherapy

INTERVENTIONS:
Radiation: Entire supraclavicular lymph node radiotherapy — Radiation is delivered to the breast/chest wall, undissected axilla, internal mammary nodes and entire supraclavicular lymph node. Entire supraclavicular lymph node includes medial supraclavicular and posterior neck lymph node.
  Arms: Breast/chest wall+undisseted axillary+IMN+entie SCL (entire SCL radiation)
Radiation: Medial supraclavicular lymph node radiotherapy — Radiation is delivered to the breast/chest wall, undissected axilla, internal mammary nodes and entire supraclavicular lymph node.
  Arms: Breast/chest wall+undisseted axillary+IMN+medial SCL ( medial SCL radiation)

SUMMARY:
Locally advanced breast cancer has high-risk local regional recurrence after surgery. Radiotherapy could reduce the local regional recurrence and improve disease free survival and overall survival. Regional lymph node irradiation is the important part of breast cancer radiotherapy. However, there are some controversies about regional lymph node delineation, especially the supraclavicular irradiation volume. Many studies had confirmed that posterolateral region of the supraclavicular fossa (also named Posterior neck lymph node) had a high risk involvement based on the mapping of recurrence nodes. This randomized phase III trial compares medial supraclavicular lymph node irradiation with entire supraclavicular lymph node irradiation in patients with pathologically positive axillary lymph node and high risk of recurrence after mastectomy or breast conservative surgery. It is not yet known if radiation works better with entire supraclavicular fossa than medial supraclavicular fossa.

DETAILED DESCRIPTION:
PRIMARY OBJIECTIVE:

I. To evaluate whether entire supraclavicular lymph node irradiation is superior to medial supraclavicular lymph node irradiation in terms of disease free survival for patients with positive lymph nodes and high risk of recurrence after breast cancer surgery

SECONDARY OBJECTIVES:

I. To estimate the difference of overall survival II. to estimate the difference of ipsilateral supraclavicular node recurrence III. to estimate the difference of local regional recurrence IV. to estimate the difference of radiation related toxicities and quality of life.

Outline: Beginning 2-12 weeks after the completion of breast cancer surgery and neoadjuvant/adjuvant chemotherapy, patients are randomized to 1 of 2 treatment arms Arm I: Patients undergo breast/chest wall, undissected axillary, internal mammary node and medial supraclavicular node radiation. Conventional fractionated radiotherapy 50Gy/25Fx/5w or hypofractionated 42.5Gy/16Fx/3.5week with IMRT or VAMT technique is recommended. 3DCRT technique is not permitted.

Arm II: Patients undergo breast/chest wall, undissected axillary, internal mammary node and entire supraclavicular node radiation. Conventional fractionated radiotherapy 50Gy/25Fx/5w or hypofractionated 42.5Gy/16Fx/3.5week with IMRT or VAMT technique is recommended. 3DCRT technique is not permitted

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0-1
2. Newly diagnosed invasive breast cancer
3. Initial clincial diagonosis stage is T1-4, N0-3a/b, M0: If neoadjuvant chemotherapy was not administered: pathological stage is T1-3N2-3a/b, M0; If neoadjuvant chemotherapy was administered：clinical stage III or pathological stage is T1-4N1-3a/bM0.
4. Underwent breast conservative surgery or Mastectomy with or without breast reconstruction with clear negative margin. At least, axillary level I and level II should be cleared with ≥10 lymph node (including the number of sentinal lymph node) . Level III dissection and internal mamamry node dissection are not required, but may be performed at the discretion of the surgeon.
5. Should receive ≥6 cycles standard neoadjuvant and/or adjuvant chemotherapy (taxane and/or anthracycline based).
6. Enrolled on the trial within 12 weeks of the later of two dates: the final breast cancer surgical procedure or administration of the last cycle of cytotoxic chemotherapy.
7. For ER and/or PR positive patients, the duration of anticipated endocrine therapy should be≥5 year ; For HER2 postive patients, the duration of anticipated herceptin should be 1 year.
8. Writtern, informed consent.

Exclusion Criteria:

1. Initinal clinical diagnosis N3c (supraclavicualr node metastasis)
2. T4 or inflamed breast cancer with no good downstage by neoadjuvant chemotherapy
3. Distant metastasis
4. Bilateral breast cancer or previously contralateral breast cancer
5. Positve sentinal lymph node with no axillary dissection
6. ECOG ≥2
7. Could not tolerate chemotherapy and anti-HER2 target treatment
8. Active infectious
9. History of radiotherapy
10. Serious medical complcation
11. Breast cancer during pregnancy and lactation
12. Had simultaneousl or previous secondary malignancies, except for skin basal cell carcinoma and cervical carcinoma in situ.
13. Inaccessibility for follow-up

    -

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS ) | Up to 5 years after completion of radiation therapy
  defined as time from randomization until to local, regional, or distant recurrence, or any death, or secondary primary cancer

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after completion of radiation therapy
  defined as time from any death
Ipsilateral supraclavicular lymph node recurrence (ISLNR) ) | Up to 5 years after completion of radiation therapy
  defined as entire ipsilateral supraclavicular lymph node recurrence
Local reigonal recurrence (LRR) | Up to 5 years after completion of radiation therapy
  chest wall, breast , regional lymph node recurrence
Distance metastasis (DS) | Up to 5 years after completion of radiation therapy
  any recurrence in all areas beyond local, regional and death due to breast cancer
incidence of adverse events | Up to 5 years after completion of radiation therapy
  Adverse events categorized using the NCI Common Terminology for Adverse Events Version 4.0 (CTCAE v4.0)
difference of quality of life | Up to 5 years after completion of radiation therapy
  evaluate the quality of life according to EROTC-QLQ-C30 and QLQ BR23
differences in upper limb function | Up to 5 years after completion of radiation therapy
  evaluate the upper limb function by Quick-dash

CONTACTS AND LOCATIONS:
Overall Officials: Zhaozhi Yang, M.D, Principal Investigator — Fudan University; Xiaomao Guo, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Mei X, Hu Z, Yu B, Zhang C, Li Y, Liu K, Ma X, Ma J, Chen X, Meng J, Shi W, Wang X, Mo M, Shao Z, Zhang Z, Yu X, Guo X, Yang Z. Adjuvant medial versus entire supraclavicular lymph node irradiation in high-risk early breast cancer (SUCLANODE): a protocol for a multicenter, randomized, open-label, phase 3 trial. BMC Cancer. 2024 Jan 9;24(1):49. doi: 10.1186/s12885-024-11831-8. PMID 38195438